CLINICAL TRIAL: NCT06695936
Title: Treatment with Intensity Modulated Radiotherapy on the Change of Cognitive Function in Nasopharyngeal Carcinoma Patients: a Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Other Study IDs: 2024-FXY-132
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Nasopharyngeal Carcinoma (NPC); Cognitive Function
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational cohort study aimed at investigating changes in hippocampal function and its impact on cognitive function in newly diagnosed nasopharyngeal carcinoma patients without metastasis, from baseline to a period after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed nasopharyngeal carcinoma patients confirmed by pathology, who have not received surgical, induction chemotherapy, radiotherapy, or other anti-tumor treatments;
* Clinical stage classified as AJCC 8th edition Stage I-IVa, with no distant metastasis, and who are scheduled to undergo intensity-modulated radiotherapy (IMRT) according to clinical plans;
* Pathologically diagnosed as non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated type, i.e., WHO type II or III);
* All participants are Han Chinese and right-handed;
* Age between 18 and 60 years, with an education level of junior high school or above;
* No history of neurological diseases or head trauma;
* No other severe systemic diseases other than nasopharyngeal carcinoma;
* No hippocampal invasion before treatment;
* Routine MRI before treatment shows no abnormal lesions in the hippocampus;
* No family history of mental illness.

Exclusion Criteria:

* Routine MRI before treatment shows abnormal lesions in the hippocampus;
* Contraindications for magnetic resonance examination;
* Concurrent other brain diseases;
* Pathologically diagnosed as keratinizing squamous cell carcinoma (WHO type I);
* Patients with recurrence or distant metastasis;
* Patients who have previously undergone radiotherapy or chemotherapy;
* Abnormal function of vital organs such as heart, brain, or lungs;
* History of head trauma or mental/neuro diseases;
* Age less than 18 years or greater than 60 years;
* Patients whose initial treatment plan is changed during the observation
* period due to disease progression (including residual tumors after
* radiotherapy, tumor recurrence, or newly developed distant metastasis);
* Patients with diabetes or hypertension;
* Those unable to cooperate in completing neurocognitive scale testing;
* Those with other uncontrolled severe diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Untreated newly diagnosed nasopharyngeal carcinoma patients without metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2028-11-15 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of cognitive decline. | 2 years
  In a cohort of nasopharyngeal carcinoma patients undergoing intensity-modulated radiotherapy, we will observe the incidence of cognitive decline from baseline, at the end of radiotherapy, and post-treatment. The study will investigate the impact of hippocampal radiation dose on cognitive function in these patients and summarize the patterns of change.

SECONDARY OUTCOMES:
The relationship between hippocampal atrophy, radiation dose, and cognitive function after radiotherapy. | 2 years
  Statistical analysis will be conducted based on the changes in hippocampal volume before and after radiotherapy, tumor target dose, hippocampal irradiation dose, and cognitive function scale test results.
The relationship between hippocampal functional impairment, radiation dose, and cognitive function after radiotherapy. | 2 years
  Using resting-state fMRI technology, individual local brain function and default network information will be obtained. Variance analysis will be used to compare hippocampal changes before and after radiotherapy, clarifying the relationship between hippocampal functional damage, radiation dose, and cognitive function post-radiotherapy.
The relationship between hippocampal microstructural damage, radiation dose, and cognitive function after radiotherapy. | 2 years
  Using Synthetic MRI imaging technology, imaging data of nasopharyngeal carcinoma patients will be collected before and after radiotherapy to provide individual whole-brain quantitative parameters and hippocampal microstructural information. Variance analysis will be used to compare pre- and post-radiotherapy differences, elucidating the relationship between hippocampal microstructural damage, radiation dose, and cognitive function.
The relationship between hippocampal microvascular injury, radiation dose, and cognitive function after radiotherapy. | 2 years
  Based on multimodal MRI technology, this study will explore the microvascular status and changes in blood perfusion in nasopharyngeal carcinoma patients before and after radiotherapy, clarifying the relationship between hippocampal microvascular damage, radiation dose, and cognitive function post-radiotherapy.
The impact of different chemoradiation treatment modalities on the occurrence of cognitive decline. | 2 years
  According to the TPS planning system dose statistics and dose-volume histogram, we will quantify the irradiation dose-volume of critical organs, including: hippocampal volume, tumor target volume, clinical target volume, and planning target volume; maximum dose and average dose of the hippocampus, as well as parameters on the dose-volume histogram. The cognitive function of patients after radiotherapy will be evaluated based on common adverse events as defined by CTCAE.
The correlation between cognitive decline after radiotherapy and quality of life. | 2 years
  "The quality of life will be prospectively assessed before treatment and followed up continuously after radiotherapy."